CLINICAL TRIAL: NCT03185507
Title: The Effect of Cryotherapy on Cerebral Hemodynamics Within Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jacob Resch, Assistant Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19706
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Cryotherapy Effect; Oxygen Deficiency
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: Thirty-four healthy participants were recruited from a large urban university. Participants were included if they were healthy and between the age of 18 and 25 years old. After obtaining consent, participants completed symptom, mood and medical history inventories. After determining if a participant met inclusion criteria, the subject remained seated at a testing station for a 10-minute rest period prior to NIRS data collection. Randomization was performed a priori using a random number generator and was stratified on sex. Participants either received superficial cryotherapy or sat quietly for 20 minutes.
Who Masked: Investigator
Masking Description: The was a randomized single-blind study. Only the clinician was blinded to which intervention was administered to each randomly assigned participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy (Experimental): Participants received superficial cryotherapy using the Cryohelmet(TM)
  Interventions: Device: CryoHelmet
- Control (No Intervention): Participants sat quietly for 20 minutes

INTERVENTIONS:
Device: CryoHelmet — Cryotherapy was administered using the Catalyst CryoHelmet™ (All-Star Sporting Goods®, Shirley, Massachusetts, USA). The CyroHelmet is a flexible helmet equipped with gel ice packs meant to cool the head and neck.
  Arms: Cryotherapy

SUMMARY:
Upon suffering a concussion, a neurometabolic cascade including an increase in glucose and oxygen demand occurs for up to 48 hours post-insult.5 This period of increased glucose and oxygen demand is coupled with a period of hyperperfusion and decreased cerebral blood flow. 6-9 Cryotherapy in the musculoskeletal system has been shown to decrease tissue temperature, blood flow, oxygen and metabolic demands.10-17 Cryotherapy following moderate or severe traumatic brain injury has been demonstrated to decrease intracranial metabolic processes and oxygenation consumption.18-23 Although the benefits of cryotherapy have been established in moderate-severe TBI, the effects of superficial cranial cooling in individuals with and without concussion are unknown. The purpose of this randomized control trial is to evaluate the effects of superficial cryotherapy on cerebral blood flow and cognitive function in healthy, recreationally active young adults.

DETAILED DESCRIPTION:
The prevalence of concussion has been estimated to be between 4,380 and 10,403 concussions per day in the United States annually with over an estimated 3 million visits to emergency departments each year.1 Symptoms following a concussion last up to 10 days for 90% of cases2; however, the reduction of symptoms in this time frame does not indicate full neurometabolic recovery.

Following concussion, a neurometabolic cascade of events immediately occurs following initial impact with return to normative values around 30 days post-injury. In an attempt to maintain homeostasis in the brain following impact, glucose and oxygen demand increases temporarily and are coupled with periods of increased hyperperfusion and decreased cerebral blood flow (CBF). Although the neurometabolic timeline immediately following impact is only generally understood, there is consensus upon acute increases in CBF and metabolic activity followed by decreased CBF until return to normative values.

Cryotherapy has been studied extensively for its' effects throughout the musculoskeletal system. Cryotherapy in the musculoskeletal system has been shown to decrease tissue temperature and blood flow, as well as decrease oxygen and energy demands.12-19 Cryotherapy has also been applied in cases of moderate or severe traumatic brain injury and has demonstrated to decrease intracranial metabolic processes and oxygenation consumption. Although the potential benefits of cryotherapy have been established in cases of moderate to severe traumatic brain injury (TBI), there is no current research examining cryotherapy in the treatment of concussion.

A convenience sample of 34 healthy, recreationally active individuals between the ages of 18-25 years will be recruited for participation in this study. The independent variable in this study will be group (cryotherapy, control). The primary outcome measures of interest are cognitive functioning measured using the Stroop Test and cerebral blood hemodynamics and hemoglobin saturation measured using near infrared spectroscopy. The pain visual analog scale (VAS) will be used to quantify tolerance to the intervention.

The following study will address the following objectives and related hypotheses:

Objective 1: To determine if the application of cryotherapy influences intracranial hemodynamics within healthy recreationally active young adults.

Hypothesis 1: Cryotherapy will cause a decrease in intracranial hemodynamics; specifically, the CO2 saturation and deoxygenated hemoglobin causing a decrease in intracranial metabolic activity.

Objective 2: To determine if the application of cryotherapy decreases cerebral blood flow within healthy recreationally active individuals.

Hypothesis 2: The application of cryotherapy will not cause a change in cerebral blood flow due to the highly regulated central nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 25 years of age
* Recreationally active (exercise at least 30 minutes, 3 times weekly)

Exclusion Criteria:

* Contraindications for cryotherapy (eg. Raynaud's phenomenon, cold urticaria)
* Any documented learning difficulty or disability
* Any known neurological or psychiatric disorder
* History of migraines
* History of a concussion or traumatic brain injury in past 6 months
* Currently taking psychotropic medications
* Any known metabolism diseases
* Any known hematological diseases
* Any recreational drug use in past month
* Any known cardiopulmonary impairments or pathologies

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
Oxygenated blood | Oxygenated blood was collected throughout the data collection period (45 minutes)
  Oxygenated blood based on functional near-infrared spectroscopy (fNIRS) data output
Deoxygenated blood | Dexoygenated blood was collected throughout the data collection period (45 minutes)
  Deoxygenated blood based on functional near-infrared spectroscopy (fNIRS)
Stroop Task reaction time | Stroop Task reaction time was collected prior to and following the intervention. Each test took approximately 5 minutes to complete.
  Reaction time measured in milliseconds while completing the Stroop Task

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia Memorial Gymnasium, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jackson K, Rubin R, Van Hoeck N, Hauert T, Lana V, Wang H. The effect of selective head-neck cooling on physiological and cognitive functions in healthy volunteers. Transl Neurosci. 2015 Jun 26;6(1):131-138. doi: 10.1515/tnsci-2015-0012. eCollection 2015. PMID 28123796